CLINICAL TRIAL: NCT05057637
Title: The Impact of Optical Coherence Tomography on the Decision-making Process of Endovascular Treatment of Femoropopliteal Disease
Brief Title: The Impact of Optical Coherence Tomography on the Endovascular Treatment Planning of Femoropopliteal Disease
Acronym: Optimo
Status: Active, not recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: Optimo study
Record Dates: First submitted 2021-09-01; First posted 2021-09-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Femoropopliteal Stenosis
Keywords: optical coherence tomography; digital subtraction angiography; endovascular treatment planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Complete cohort: In all patients included in the study subsequent optical coherence tomography (OCT) measurements will be performed pre and post stent placement.
  Interventions: Device: Optical coherence tomography measurements

INTERVENTIONS:
Device: Optical coherence tomography measurements — Optical coherence tomography measurements in femoropopliteal tract
  Other Names: Ilumien Optis

SUMMARY:
Rationale: Peripheral arterial disease is a severe clinical problem with an increasing prevalence, due to an ageing population. Endovascular treatment, usually using stents, is recommended for most lesions in the femoropopliteal tract. The patency of these stents is influenced by several factors, including stent sizing and stent positioning.

Current procedural planning of femoropopliteal disease is primarily based on single-plane digital subtraction angiographies (DSA). This modality provides a 2-dimensional image of the vessel lumen, which may be suboptimal for stent sizing. It can therefore be difficult to choose the optimal stent position as minor lesions may be missed. Suboptimal treatment could result in unfavourable levels of wall shear stress causing the vessel wall to be more susceptible to neo-intimal hyperplasia ultimately causing restenosis and stent failure. Intravascular optical coherence tomography (OCT) is able to visualize the arterial wall with a micrometer resolution, which could result in better stent sizing. Furthermore, OCT is able to visualize different layers in the vessel wall and identify unhealthy areas, which may lead to a more optimal stent placement as unhealthy areas can be covered completely. Moreover, OCT provides detailed patient-specific geometries necessary to develop reliable computational fluid dynamics (CFD) models that simulate blood flow in stented arteries and calculate wall shear stresses, which could predict stent patency.

Objective: To investigate in a clinical study how often the use of intravascular optical coherence tomography for femoropopliteal stenotic lesions leads to alterations in treatment planning before and after stent placement, in comparison to traditional digital subtraction angiography-based treatment planning.

Study design: Exploratory observational study. Study population: 25 patients with femoropopliteal stenotic lesions who are treated with a Supera interwoven nitinol stent or Absolute nitinol stent.

Main study parameters/endpoints: The percentage of procedures in which OCT changed the DSA-based treatment planning before and after stent placement to investigate the impact of OCT imaging on treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of older
* Written informed consent
* Scheduled endovascular treatment of femoropopliteal stenotic lesions with a Supera interwoven nitinol stent or Absolute nitinol stent
* Clinically and hemodynamically stable

Exclusion Criteria:

* Occluded superficial femoral artery or popliteal artery
* Superficial femoral artery and/or popliteal artery diameter larger than 6.5 mm
* Severely impaired renal function (eGFR < 30 ml/min), end stage renal disease
* Cardiac insufficiency (NYHA 3-4)
* Hypersensitivity to iodinated contrast media
* BMI > 25 and contralateral approach not possible
* Minimal lumen diameter of target lesion < 1.5 mm
* Presence of a hemodynamically significant inflow stenosis in the aorto-iliac tract or the common femoral artery
* Participating in another trial with an investigational drug or medical device concerning the femoropopliteal tract interfering with the current study
* Life expectancy of less than 24 months
* Women of child-bearing age not on active birth control
* Legally incapable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with one or more stenotic lesions in the femoropopliteal tract that are scheduled for endovascular treatment with a Supera interwoven nitonol stent or Absolute nitinol stent.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Changed treatment planning based on OCT | Immediately following the procedure
  The percentage of procedures in which the OCT changed the DSA-based treatment planning before and after stent placement to investigate the impact of OCT imaging on treatment planning.

SECONDARY OUTCOMES:
Presence of artefacts in CTA scan | 6-8 weeks after the procedure
  The presence of artefacts will be used to determine the image quality of the CTA scan
Presence of artefacts in OCT scan | Immediately following the procedure
  The presence of artefacts will be used to determine the image quality of the OCT scan
Segmented vessel lumen based on CTA scan | Up to 2 years after the procedure
  The vessel lumen in the CTA scan will be segmented to obtain a patient-specific geometry.
Segmented vessel lumen based on OCT scan | Up to 2 years after the procedure
  The vessel lumen in the OCT scan will be segmented to obtain a patient-specific geometry.
Correlation CTA-based and OCT-based vessel lumen segmentations | Up to 2 years after the procedure
  The obtained CTA-based segmentation will be compared to the OCT-based segmentation. The vessel radius along the blood vessel for both the CTA-based and OCT-based segmentation will be compared point-by-point after which the correlation beteen both segmentations will be obtained
Velocity streamlines obtained from CTA-based CFD simulation | Up to 2 years after the procedure
  Velocity streamlines are calculated using a computational fluid dynamics model based on the CTA-based vessel lumen segmentation.
Time averaged wall shear stress obtained from CTA-based CFD simulation | Up to 2 years after the procedure
  The second parameter calculated using the CTA-based CFD simulation is the time averaged wall shear stress. This is the wall shear stress averagerd over one heartbeat.
Velocity streamlines obtained from OCT-based CFD simulation | Up to 2 years after the procedure
  Velocity streamlines are calculated using a computational fluid dynamics model based on the OCT-based vessel lumen segmentation.
Time averaged wall shear stress obtained from OCT-based CFD simulation | Up to 2 years after the procedure
  The second parameter calculated using the OCT-based CFD simulation is the time averaged wall shear stress. This is the wall shear stress averagerd over one heartbeat.
Late luminal loss | Up to 2 years after the procedure
  Defined as the vessel diameter right after procedure minus the vessel diameter during follow-up
Correlation between late luminal loss and CTA-based CFD | Up to 2 years after the procedure
  The regions with late luminal loss will be compared to regions with disturbed velocity streamlines and low time averaged wall shear stress (<0.4 Pa) calculated with the CTA-based CFD. This correlation shows how well the CTA-based CFD model can predict late luminal loss.
Correlation between late luminal loss and OCT-based CFD | Up to 2 years after the procedure
  The regions with late luminal loss will be compared to regions with disturbed velocity streamlines and low time averaged wall shear stress (<0.4 Pa) calculated with the OCT-based CFD. This correlation shows how well the OCT-based CFD model can predict late luminal loss.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, prof, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No